CLINICAL TRIAL: NCT06677593
Title: Detection of Electrodermal Activity in Pain (DEEP)
Brief Title: Detection of Electrodermal Activity in Pain 2
Acronym: DEEP 2
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Skov Benthien, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-24037808-Phase-2
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Chronic Obstructive Pulmonary Disease (COPD; Pain
Keywords: pain; electrodermal activity; pain detection; pain prediction; galvanic skin response; wearable; pain monitoring
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients with COPD or cancer

SUMMARY:
The goal of this study is to investigate the association between self-reported pain and electrodermal activity and to create an algorithm that detects pain and provides timely alarms for rising pain levels in patients with life-threatening illnesses suffering from persistent pain. The study is exploratory.

Hypothesis: Electrodermal activity can distinguish different pain intensity levels in patients with chronic pain and a life-threatening disease.

Methodology: Thirty-seven patients with cancer and/or chronic obstructive pulmonary disease (COPD) will be identified through hospital record screening. These patients will wear a monitoring device for a maximum of one week and report their pain intensity throughout the day.

Analysis: Discriminant analysis will be used to differentiate between mild, moderate, and severe pain. This study is exploratory, generating hypotheses for subsequent phases of the project.

DETAILED DESCRIPTION:
Methods The study is a phase 2 trial, preceded by a phase 1 trial that included healthy volunteers.

Patients will be inpatients and outpatients at Department of Pulmonary and Endocrine Diseases, Hvidovre Hospital.

Measures Subjective measures (self reported) Pain. Pain intensity (interval, 0 to 10) is measured using the NRS, a commonly used tool asking patients to rate their pain intensity on a scale from 0 to 10, with 0 indicating no pain and 10 reflecting the worst possible pain.

Patient Health Status. The Patient Health Questionnaire (PHQ-9) is used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings. The PHQ-9 is the depression module.

Ambulatory assessment. The patient group in phase 2 will be asked to wear a wristband device for 1 week. During this period, a prompt will be sent on a smartphone connected to a wearable device provided by Movisens GmbH, five times a day (9 am, 12 pm, 3 pm, 6 pm, and 9 pm) to answer questions about their current pain levels using the NRS scale.

Objective measures Electrodermal activity. A wearable device provided by Movisens GmbH will be used to record skin conductance measured in microsiemens (μS).

Wearable device The EdaMove 4 device provided by Movisens GmbH consists of an EDA and activity sensor. It records EDA signals to monitor both tonic and phasic electrical activity in the skin.

ELIGIBILITY:
Inclusion Criteria:

* Danish
* Age over 18
* Persistent or recurrent pain (longer than three months)
* Cancer: DC01-DC9 or Pulmonary Diseases:DJ40-DJ47

Exclusion Criteria:

* A current diagnosis with psychological/ psychiatric disorders
* Impaired cognitive function
* Substance abuse
* A skin condition on the to-be-tested body parts
* PHQ-9 reveals suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hvidovre Hospital
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | while participants wear the device (up to 7 days)
  Numerical rating scale score. Pain intensity (interval, 0 to 10) is measured using the NRS, a commonly used tool asking patients to rate their pain intensity on a scale from 0 to 10, with 0 indicating no pain and 10 reflecting the worst possible pain.

SECONDARY OUTCOMES:
Skin conductance level | while participants wear the device (up to 7 days)
  The average skin conductance value (μS) for 10 seconds.
Number of Skin Conductance Fluctuations | while participants wear the device (up to 7 days)
  Peaks with minimum amplitudes of 0.02 μS and a slope rate < 2 μS/s, in 10 second intervals
Patient Health Questionnaire (PHQ-9) | administered the day of enrollment
  The Patient Health Questionnaire (PHQ-9) will be used to screen participants as symptoms of depression in order to control during the statistical analysis.
  The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day), providing a 0 to 27 severity score.
Pain frequency | while participants wear the device (up to a period of 7 days)
  Number of patient reported pain episodes of pain intensity over 5 (using the NRS pain intensity scale)
Pain evaluation from healthcare personale not possible | in the duration that the participant wears the device (up to 7 days)
  Evaluate how often it is not possible to estimate pain levels for patients, thus, a need for a tool to assist). This is marked at the patient journal.
Medication list | while participants wear the device (up to 7 days)
  The list of medication a participant takes on regular basis during the week they will be assessed. This data will be collected from the patient journals to control and to understand the final dataset.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine S Benthien, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Copenhagen University Hospital - Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No